CLINICAL TRIAL: NCT04457414
Title: Learning Curve of Inexperienced Trainees for Identifying Cricothyroid Membrane With Ultrasound in Pediatric Patients
Brief Title: Identifying Cricothyroid Membrane With Ultrasound
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: 2005-230-113
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cannot-intubate cannot-ventilate situations in healthy children are uncommon but are often associated with poor outcome. We studied the learning curves of inexperienced trainees for identifying cricothyroid membrane with ultrasound in pediatric patients. After watching an instructional video, 30 trainees performed 5 cricothyroid membrane identification on pediatric patients undergoing general anesthesia. We analysed their learning curves relative to performance time and ultrasound anatomy of cricothyroid membrane and relative structures.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing general anesthesia

Exclusion Criteria:

* previous history of tracheostomy
* previous history of operation on neck

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients undergoing general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Performance time for identifying cricothyroid membrane with ultrasound | from immediately after anesthetic induction to end of surgery

SECONDARY OUTCOMES:
ultrasound anatomy of cricothyroid membrane | from immediately after anesthetic induction to end of surgery
  depth from skin surface, thickness, diameter, relative vessels

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea